CLINICAL TRIAL: NCT01399528
Title: A Pharmacogenomic Exploration of Lacosamide Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: St. James's Hospital, Ireland (Other); University College, London (Other); Erasme University Hospital (Other); Duke University (Other)
Responsible Party: Principal Investigator, Norman Delanty, Consultant Neurologist, Royal College of Surgeons, Ireland
Other Study IDs: RCSI_LCM
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Collecting DNA from blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Beaumont Hospital, Dublin, Ireland
- St. James' Hospital, Dublin, Ireland
- Hôpital Erasme, Brussels, Belgium
- Duke Medical Centre, North Carolina, USA
- The Institute of Neurology/University College London, UK

SUMMARY:
This is an observational study exploring the genetics of lacosamide response. The study will last 3 years and has been divided in to three stages; 1) recruitment, 2) observational phase, 3) genotyping and analysis. Patients initiating lacosamide are recruited and their baseline seizure frequency is assessed retrospectively. Patients are then monitored for 18 months with an assessment (via interview and where possible seizure diaries) of seizure frequency and other treatment related phenotypes every 3 months. The recruitment period will span months 1-12, the observational period will span months 1-30 and analysis of data will be conducted between months 30-36 (see Figure 2 below). Target sample size is 610.

Primary objective: To determine the clinical relevance of genetic variation in predicting lacosamide responsive and non-responsive patients.

Secondary objectives: To determine the clinical relevance of genetic variation in predicting:

* Optimal dose of lacosamide
* Adverse drug reactions to lacosamide

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with partial onset seizures (simple and/or complex) with or without secondary generalization (based on 1981 ILAE seizure classification scheme)
* Over 18 and under 65 years of age at date of recruitment in to the study
* Currently undergoing pharmacological treatment for refractory partial epilepsy ('refractory' here refers to patients who continue to have seizures despite treatment (current) with two or more appropriate anti-epileptic drugs at appropriate doses)
* Deemed suitable for treatment with lacosamide (following drug guidelines)

Exclusion Criteria:

* Patients experiencing seizure type other than partial onset seizures (with/without secondary generalisation)
* Patients with a history of chronic alcohol or drug abuse within previous 3 years.
* Non refractory epilepsy patients
* Patients suffering any other clinically significant disease e.g. cancers, progressive neurological disorder, heart failure, respiratory failure etc
* Patients who are pregnant or who are intending on getting pregnant within the period of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with epilepsy recruited from five tertiary referral centres.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | Recorded daily by participant. Passed on to study researchers every 3 months for an 18 month period
  We will record seizure type and frequency. Seizure types will follow definitions as provided by the International League Against Epilepsy. Seizure frequency will be as recorded by the participant in a seizure diary.

SECONDARY OUTCOMES:
Maintenance dose | Recorded every three months for an 18 month period
  Maintenance dose will be defined as the tolerated daily dose required by the patient for seizure control.
Adverse drug reactions | Recorded as reaction arise during the 18 month study period
  We will record any adverse reactions recorded by the study participant, including for example (but not limited to): dizziness, ataxia, vomiting, diplopia, nausea, vertigo, and vision blurred.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Delanty, MB FRCPI, Principal Investigator — Beaumont Hospital and Royal College of Surgeons in Ireland; Gianpiero L Cavalleri, PhD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (5):
- Duke Medical Centre, Durham, North Carolina, United States
- Hospital Erasme, Brussels, Belgium
- Ireland (2):
  - Beaumont Hospital, Dublin, Dublin
  - St.James Hospital, Dublin
- The Institute of Neurology, London, United Kingdom